CLINICAL TRIAL: NCT04451187
Title: A Multicentric, Randomized, Double-Blind, Placebo- and Positive-Controlled 4-way Crossover Study to Evaluate the Effects of Single and Repeated Administration of Oral Seltorexant as an add-on Medication to an Antidepressant on On-Road Driving Performance in Participants With Major Depressive Disorder
Brief Title: A Study of Oral Seltorexant as an add-on Medication to an Antidepressant on On-road Driving Performance in Participants With Major Depressive Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CR108762; 42847922MDD1005 (Other: Janssen Research & Development, LLC); 2019-004913-15 (EudraCT Number)
Record Dates: First submitted 2020-06-26; First posted 2020-06-30 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant; zopiclone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment Sequence CADB (Experimental): Participants will receive placebo once daily (OD) at bedtime for 8 consecutive days from Day 1 to Day 8 (Treatment C) in Period 1 followed by Dose 1 of seltorexant tablets and placebo OD at bedtime for 8 consecutive days from Day 1 to Day 8 (Treatment A) in Period 2 followed by Dose 2 of seltorexant tablets OD at bedtime for 8 consecutive days from Day 1 to Day 8 (Treatment D) in Period 3 followed by zopiclone on Day 1 and Day 8 and placebo from Day 2 to Day 7 OD at bedtime (Treatment B) in Period 4. There will be a washout period of 5 to 21 days between each period.
  Interventions: Drug: Seltorexant Dose 1; Drug: Seltorexant Dose 2; Drug: Placebo; Drug: Zopiclone
- Treatment Sequence ABCD (Experimental): Participants will receive Treatment A in Period 1 followed by Treatment B in Period 2 followed by Treatment C in Period 3 followed by Treatment D in Period 4. There will be a washout period of 5 to 21 days between each period.
  Interventions: Drug: Seltorexant Dose 1; Drug: Seltorexant Dose 2; Drug: Placebo; Drug: Zopiclone
- Treatment Sequence BDAC (Experimental): Participants will receive Treatment B in Period 1 followed by Treatment D in Period 2 followed by Treatment A in Period 3 followed by Treatment C in Period 4. There will be a washout period of 5 to 21 days between each period.
  Interventions: Drug: Seltorexant Dose 1; Drug: Seltorexant Dose 2; Drug: Placebo; Drug: Zopiclone
- Treatment Sequence DCBA (Experimental): Participants will receive Treatment D in Period 1 followed by Treatment C in Period 2 followed by Treatment B in Period 3 followed by Treatment A in Period 4. There will be a washout period of 5 to 21 days between each period.
  Interventions: Drug: Seltorexant Dose 1; Drug: Seltorexant Dose 2; Drug: Placebo; Drug: Zopiclone

INTERVENTIONS:
Drug: Seltorexant Dose 1 — Participants will receive Dose 1 of seltorexant OD from Day 1 to Day 8 as part of Treatment A as per assigned treatment sequence.
  Other Names: JNJ-42847922
Drug: Seltorexant Dose 2 — Participants will receive Dose 2 of seltorexant OD from Day 1 to Day 8 as part of Treatment D as per assigned treatment sequence.
  Other Names: JNJ-42847922
Drug: Placebo — Participants will receive placebo of seltorexant OD from Day 1 to Day 8 as a part of Treatment A and C and from Day 2 and Day 7 as a part of Treatment B as per assigned treatment sequence.
Drug: Zopiclone — Participants will receive Dose 3 of zopiclone OD from Day 1 to Day 8 as a part of Treatment B as per assigned treatment sequence.

SUMMARY:
The purpose of the study is to evaluate the effect of seltorexant, compared to placebo, as an add-on medication to an antidepressant, on next-day driving performance as assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test in participants with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Participant with major depressive disorder (MDD) (not applicable for elderly without MDD) must meet Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) diagnostic criteria for major depressive disorder (MDD) without psychotic features based upon clinical assessment (DSM-5 296.20, 296.21, 296.25, 296.26, 296.30, 296.31, 296.35 or 296.36) and confirmed by the Mini International Neuropsychiatric Interview (MINI) and the attending general physician, psychiatrist or mental health practitioner. The MINI will also be conducted for elderly participants without MDD to rule out major psychiatric disorders
* Participants with MDD (not applicable for elderly without MDD) must have mild or better depressive symptoms indicated by a Montgomery-Asberg Depression Rating Scale (MADRS) total score of less than or equal to (<=) 18 at screening
* Participants with MDD having comorbid generalized anxiety disorder, social anxiety disorder, or panic disorder for whom major depressive disorder (MDD) is considered the primary diagnosis are not excluded
* Participants with MDD (not applicable for elderly without MDD) must be receiving and tolerating well any one of the following selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for depressive symptoms in any formulation and available in the participating country: citalopram, duloxetine, escitalopram, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine at a stable dose (at therapeutic dose level) for at least 4 weeks prior to screening, and expected to continue to take the same drug and dose for the duration of the study
* Participant should be medically stable on the basis of medical history, neurological examination and clinical laboratory tests performed at screening, and physical examination, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and predose on Day 1 of Period 1.

Exclusion Criteria:

* Participants has a recent (last 3 months) history of, or current signs and symptoms of severe renal insufficiency (creatinine clearance less than [<]30 milliliter per minute [mL/min]); clinically significant or unstable cardiovascular, respiratory, gastrointestinal, neurologic, hematologic, rheumatologic, immunologic or endocrine disorders; and participants with uncontrolled type 1 or type 2 diabetes mellitus
* Participants has clinically significant hepatic disease as defined by greater than or equal to (>=) 2* Upper Limit of Normal [ULN]) increase of aspartate aminotransferase (AST) or alanine aminotransferase (ALT) at screening (one retest is permitted); and significant liver disease including cirrhosis, ascites, active hepatitis etc. (fatty liver disease or Gilbert's syndrome will be allowed as long as it does not meet the above criteria)
* Participants has current signs/symptoms of hypothyroidism or hyperthyroidism. For participants with a history of thyroid disease and for participants who, regardless of thyroid history have the thyroid stimulating hormone (TSH) value out of range, a free thyroxine (FT4) test will be conducted. If the FT4 value is abnormal and considered to be clinically significant (after discussion with the medical monitor) the participant is not eligible. Participants with a pre-existing history of thyroid disease/disorder who are treated with thyroid hormones need to be on a stable dosage for 3 months prior to the start of the screening phase. Participants taking thyroid supplementation for antidepressant purposes are not allowed in the study
* Participants has Cushing's Disease, Addison's Disease, primary amenorrhea, or other evidence of significant medical disorders of the hypothalamic-pituitary-adrenal (HPA) axis
* Participants has a lifetime history of narcolepsy and seizures (except childhood seizures)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

PRIMARY OUTCOMES:
Driving Performance as Assessed by the Mean Difference of SDLP From an on-road Driving Test | Day 2
  In the participants with major depressive disorder (MDD), driving performance will be assessed by the mean difference of standard deviation of lateral position (SDLP) from an on-road driving test to evaluate the effect of seltorexant dose 1, compared to placebo, as an add-on medication to an antidepressant.
Driving Performance as Assessed by the Mean Difference of SDLP From an on-road Driving Test | Day 9
  In the participants with MDD, driving performance will be assessed by the mean difference of SDLP from an on-road driving test to evaluate the effect of seltorexant dose 1, compared to placebo, as an add-on medication to an antidepressant.

SECONDARY OUTCOMES:
Driving Performance as Assessed by the Mean Difference of SDLP From an on-road Driving Test | Day 2 and Day 9
  The driving performance will be assessed by the mean difference of SDLP from an on-road driving test to evaluate the effect of seltorexant doses (Dose 1 and Dose 2), compared to placebo in adult participants with major depressive disorder (MDD); and on adults and elderly participants with MDD and healthy elderly (if enrolled) (seltorexant Dose 1 and Dose 2); and on adults and elderly participants with MDD (seltorexant Dose 2).
Participant Driving Performance as Assessed by Visual Analog Scale | Day 2 and Day 9
  Immediately after each driving test, participants with MDD or in healthy elderly participants (if enrolled) will indicate the perceived quality of their driving performance on a visual analog scale from 0 ('I drove exceptionally poorly') to 20 ('I drove exceptionally well') around a midpoint of 'I drove normally'.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to 20 weeks
  An adverse event is any untoward medical occurrence in a clinical study participant with MDD or in healthy elderly participants (if enrolled) administered a medicinal (investigational or non investigational) product. An adverse event does not necessarily have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non investigational) product, whether or not related to that medicinal (investigational or non investigational) product.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (2):
- Anima, Alken, Belgium
- Universitaetsklinikum der RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency